CLINICAL TRIAL: NCT00524394
Title: Characteristics of Cord Blood Immunologic Parameters of Infants < 32 Weeks Gestation
Brief Title: Characteristics of Cord Blood Immunologic Parameters of Infants <32 Weeks Gestation
Acronym: AOS
Status: Terminated | Type: Observational
Why Stopped: recruitment not possible
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Other Study IDs: HSC-MS-07-0021
Record Dates: First submitted 2007-08-30; First posted 2007-09-03 (Estimated); Results first posted 2015-12-14 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-11

CONDITIONS: Premature Birth; Sepsis
Keywords: VLBW; sepsis; diagnosis; suspected sepsis
MeSH Terms: conditions — Premature Birth; Sepsis; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum only
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Infants in the NICU are at high risk for morbidity and mortality from infections of any onset. Diagnosis of these infections is imperfect at best. Patterns of inflammatory and regulatory proteins (cytokines & chemokines, in addition to antigen detection on antibody secreting cells (ASC's)may provide a more accurate and rapid approach to diagnosis of infections in these high-risk patients.

DETAILED DESCRIPTION:
Sampling methods/Data collection

Samples: Serum (1-2ml) from enrolled infants will be collected from cord blood (T0). Serial samples (0.5-1ml) will be collected at 3 other times: T1= 4-7 days, T2=10-14 days, T3= 20-30 days. These can be drawn at initiation of any sepsis work-up, or prior to any transfusion of PRBC's or when any blood ≥0.5ml will be wasted. These collections are intended to analyze the immunologic milieu in infants at various stages of natal and post-natal immune adaptation:

1. baseline levels from a relatively privileged environment (cord blood T0)
2. peak of immunogenic response after prenatal exposure (T1)
3. plateau of immunogenic response after perinatal exposure (T2)
4. relative state of equilibrium with surrounding flora (T3)

Data collection:

Baseline statistics at enrollment: Birth weight, obstetrical assessment of gestational age, mode of delivery, presence of labor, presence of IAI, ROM, intrapartum antibiotics type and length, With each sampling, data will be gathered via chart review on each infant. We will also gather data at 60 DOL, discharge, or death on any infant enrolled.

Measurements:

Experimental laboratory:

Cytokines- Each sample will have plasma analyzed by Luminex (Biorad) to determine profiles of cytokines: IL-2, IL-6, IL-8, IL-13, MIP1b, MCP1, IL-1b, IL-4, IL-5, IL-7, IL-10, IL-12p70, IL-17, GMCSF, IFN-gamma, and TNF-alpha. Standard curves for each cytokine measurement were run to determine upper and lower limits of detection.

ASC- will be quantified by enzyme-linked immunospot assay (ELISPOT) for specific isotypes IgA, IgM, and IgG. They will also be linked to 3 particular immunogenic agents: GBS, Candida, and CoNS.

Clinical laboratory:

Total WBC and band ratio will be run in the routine course of care for these infants. This is not an additional sample.

serious bacterial infections other than sepsis (meningitis, UTI)

* Course of Study- 0-30 days of life for sampling. 0-60 days of life for data collection.
* Enrollment- consecutive admissions of NICU under the following criteria

Inclusion:

Admitted to NICU at MHCH

* 1500gm or ≤ 32 wk GA Birth to <31 days of life at time of enrollment

Exclusion:

Known or suspected immunodeficiency (including maternal HIV or other known congenital infection) Known major congenital anomaly

* Recruitment Will include each eligible infant by the primary investigator or co-investigators. Assuming an incidence of LOS of ~25% and EOS of ~1-3%, a power of 80%, we should enroll 50 infants. This coincides with prior studies evaluating ASC's response in neonates, and those evaluating cytokines in cord blood and post-natally.
* Known Risks There will be no additional blood draws. There will be collection of a greater volume of blood (additional 0.5ml-1.0ml depending on size of infant) during clinical indications for blood draws. No clinical decisions will be made based on the data obtained.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at Children's Memorial Hermann Hospital with cord blood available < 1500gm or < 32 weeks gestation by OB estimate

Exclusion Criteria:

* Outborn infants transferred to CMHH without cord blood available
* Parents to not consent
* > 1500gm or > 32 weeks gestation by OB estimate

Max Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature infants
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2007-08; Primary Completion 2011-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James R Murphy, PhD, Principal Investigator — University of Texas at Houston
Locations (1):
- Children's Memorial Hermann Hospital, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment using NICU ADMISSION LIST.
Groups:
- Infants 0 to 3 Days of Life >1500 g or >32 Weeks GA: Infants born at >32 weeks of gestagional age or > 1500gm between 0 to 3 Days of Life
Period: Overall Study
Arm/Group | Infants 0 to 3 Days of Life >1500 g or >32 Weeks GA
Started | 2
Completed | 1
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- INFANTS: INFANTS 0 to 3 days of life >1500 G OR >32 WEEKS GA
Arm/Group | INFANTS
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Immunological Homeostasis
Description: Describe changes in immunological homeostasis that indicate the "normal" function vs. presence of sepsis in newborn infants of various gestational ages
Time Frame: 0 to 30 days of life.
Reporting Status: Not Posted

2. Primary Outcome: Cytokines
Description: IL2 IL6 IL8 IL13 MIP1B MCP1 IL1B IL4 IL5 IL7 IL10 IL12P70 Measure of Cytokines presence and level .
Time Frame: O TO 30 DAYS OF LIFE
Population: zero participant analyzed
Groups:
- INFANTS 0 to 3 Days of Life (DOL) >1500 G OR >32 WEEKS GA: INFANTS 0 to 3 days of life born with >1500 gm OR >32 WEEKS gestational age
Arm/Group | INFANTS 0 to 3 Days of Life (DOL) >1500 G OR >32 WEEKS GA
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From begining to the end of the study period.
Groups:
- Infants0-3 Days of Life >1500g or >32 Weeks GA: Infants born at 32 weeks of gestacional age or >1500 mg at 0-3 days of life .
Arm/Group | Infants0-3 Days of Life >1500g or >32 Weeks GA
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No